CLINICAL TRIAL: NCT00721682
Title: Evaluation of Acute Pain in Maltreated Children : a Prospective, Multicentric and Controlled Study
Brief Title: Evaluation of Acute Pain in Maltreated Children
Acronym: ANTALPED
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD 08/6-K
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Pain
Keywords: Pediatry; Ill-treatment; Pain; maltreated children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: The CASE group will be composed of children for whom the medical team will have chosen to carry out a sign of alert of ill-treatment during his hospitalization and with no plausible cause of traumatism
- control: The Control group will be composed of children, consulting with the emergency care for traumatism, not having a sign of alarm and having a plausible cause of traumatism.

SUMMARY:
The hypothesis of this study is nonrecognition by the medical team of pain in maltreated children. These children would have a particular painful behaviour, "quiet". The management of their pain would be then unsuited, which could explain their complex relation with the pain in the adulthood. A pilot study realized in the CHU of Nantes on 11 files of maltreated children showed that they had very low scores of evaluation of the pain, in spite of severe traumatisms. There is, at the moment, no data in the literature on the acute pain of the maltreated children.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 6 years
* Consultation in the emergency cares for traumatism with type of fracture and/or burn
* Time of the traumatism lower than 24 hours
* Information of the two parents or the parental authority and collection of the non-opposition.

Exclusion Criteria:

* Old superior at 6 years
* Any type of traumatism other than a fracture and/or a burn
* Traumatism without possible dating or with a time of consultation higher than 24 hours
* Opposition of the parents formulated after their information by the medical team
* Child who can not have an evaluation of the pain with the chosen scales

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: maltreated children who consult in paediatric emergencies for recent fracture or burn
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The principal judgement criterion is the proportion of children without recognized pain, measured with the rating scales validated in paediatrics, in T0, in the two populations of children (maltreated and others). | 3 years

SECONDARY OUTCOMES:
Comparison of the quantitative scores of evaluation of the pain enters the two populations of children (maltreated and others) | 3 years
Agreement between the evaluations of the pain made by the nursery nurses and those done by the doctors | 3 years
Study of the correlation enters the managed painful treatments and the recommendations of painful treatment for each pathology. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Georges PICHEROT, MD, Principal Investigator — Nantes University Hospital
Locations (7):
- France (7):
  - nantes University Hospital, Nantes, Pays de la Loire Region
  - Angers university Hospital, Angers
  - Ch Cholet, Cholet
  - CHD les oudairies, La Roche-sur-Yon
  - GHH, Le Havre
  - rennes university Hospital, Rennes
  - CH Saint Nazaire, Saint-Nazaire

REFERENCES:
- [Derived] Drouineau MH, Guenego E, Sebille-Rivain V, Vrignaud B, Balencon M, Blanchais T, Levieux K, Vabres N, Picherot G, Guen CG. Do abused young children feel less pain? Child Abuse Negl. 2017 Mar;65:248-254. doi: 10.1016/j.chiabu.2017.02.002. Epub 2017 Feb 11. PMID 28196343